CLINICAL TRIAL: NCT02446730
Title: A Prospective, Multicenter, Randomized, Open-label Trial to Evaluate Efficacy and Safety of 5mg Maintenance Dose of Prasugrel in Patients With Acute Coronary Syndrome Who Underwent Percutaneous Coronary Intervention With BiomatrixTM Stent
Brief Title: Efficacy and Safety of BiomatrixTM Stent and 5mg-Maintenance Dose of Prasugrel in Patients With Acute Coronary Syndrome
Acronym: BEAUTY-II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Myung Ho Jeong, MD, PhD, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEAUTY-II
Record Dates: First submitted 2015-05-06; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Cardiac Death; Hemorrhage; Cerebrovascular Accident; Myocardial Infarction
MeSH Terms: conditions — Death; Hemorrhage; Stroke; Myocardial Infarction | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BES with Prasugel 5mg (Active Comparator): Biolimus-eluting stent with Prasugrel 5mg once daily MD
  Interventions: Device: BES (biodegradable polymer biolimus-eluting stent); Drug: Prasugel
- BES with Clopidogrel 75mg (Active Comparator): Biolimus-eluting stent with Clopidogrel 75mg once daily MD
  Interventions: Device: BES (biodegradable polymer biolimus-eluting stent); Drug: Clopidogrel

INTERVENTIONS:
Device: BES (biodegradable polymer biolimus-eluting stent) — BES implantation
  Other Names: BiomatirxTM; Biomatrix FlexTM
Drug: Prasugel
  Arms: BES with Prasugel 5mg
Drug: Clopidogrel
  Arms: BES with Clopidogrel 75mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 5mg maintenance dose (MD) of prasugrel in patients with acute myocardial infarction (AMI) who underwent percutaneous coronary intervention (PCI) with BiomatrixTM stent.

DETAILED DESCRIPTION:
About 1400 patients derived from Korean patients with acute coronary syndrome (ACS) receiving percutaneous coronary intervention (PCI) with BES(Biolimus-eluting stent, BiomatrixTM) in a routine manner will be enrolled in the investigators trial.

These patients will be randomized 1:1 to either prasugrel 5mg once daily MD or clopidogrel 75mg once daily MD after successful PCI with BES .

The investigators excluded the patients with age ≥75 years, body weight <60 kg, or history of TIA (transient ischemic attack) or stroke. Follow-up data will be collected until 1-year after index procedure.

Primary efficacy end-point defined as the composite of cardiac death, non-fatal MI, stent thrombosis and ischemic driven target vessel revascularization and safety end-points as BARC (the Bleeding Academic Research Consortium) type ≥ 2 bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can undergo percutaneous coronary intervention with Biomatrix stent with no history of TIA or stroke,
* 75 years old or younger,
* body weight of 60 kg or more and diagnosed with acute coronary syndrome

Exclusion Criteria:

* Patients with history of TIA or stroke,
* 75 years old or older,
* body weight of 60 kg or under,
* hypersensitivity to or contraindicated for heparin, aspirin, clopidogrel, prasugrel or contrast media

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
A compoiste of cardiac death, non-fatal myocardiac infarction and stroke | within the 1 year after BIOMATRIXTM Stent implantation

SECONDARY OUTCOMES:
All-cause death | within the 1 year after BIOMATRIXTM Stent implantation
Cardiac death | within the 1 year after BIOMATRIXTM Stent implantation
non-fatal myocardial infarction | within the 1 year after BIOMATRIXTM Stent implantation
Stroke | within the 1 year after BIOMATRIXTM Stent implantation
Target lesion revascularization | within the 1 year after BIOMATRIXTM Stent implantation
stent thrombosis | within the 1 year after BIOMATRIXTM Stent implantation
BARC bleeding 2,3,and 5 | within the 1 year after BIOMATRIXTM Stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Myung Ho Jeong, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Jung-Me Lee, Pusan, South Korea